CLINICAL TRIAL: NCT01317030
Title: Tear Evaluation Between Habitual Contact Lens Wearers and Non Contact Lens Wearers Using a Schirmer Strip for Tear Collection
Brief Title: Tear Evaluation Between Habitual Contact Lens Wearers and Non Contact Lens Wearers
Status: Terminated | Type: Observational
Why Stopped: Study was terminated due to a business decision to cancel the entire project.
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: ROC2-10-110
Record Dates: First submitted 2011-03-09; First posted 2011-03-17 (Estimated); Results first posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Contact Lenses, Extended-Wear

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Contact Lens Wear: Senofilcon A Lenses, using Sensitive Eyes Saline Solution and/or Biotrue Multipurpose Solution
  Interventions: Device: Contact Lens Wear
- Non-Contact Lens Wear
  Interventions: Other: Non-Contact Lens Wear

INTERVENTIONS:
Device: Contact Lens Wear — Senofilcon A lenses will be rubbed and rinsed with Bausch + Lomb Sensitive Eyes Saline. The lenses will then be placed into Biotrue multi-purpose solution and soaked for at least 10 hours but no more than 24 hours prior to lens insertion into one eye.
  Groups: Contact Lens Wear
Device: Contact Lens Wear — Senofilcon A lenses will be rubbed and rinsed each side with Bausch + Lomb Sensitive Eyes Saline just prior to lens insertion into fellow eye.
  Groups: Contact Lens Wear
Other: Non-Contact Lens Wear — No intervention
  Groups: Non-Contact Lens Wear

SUMMARY:
to evaluate tears between habitual contact lens wearers and non contact lens wearers

DETAILED DESCRIPTION:
The objective of this study is to evaluate tears between habitual contact lens wearers and non contact lens wearers using a Schirmer Strip for tear collection.

ELIGIBILITY:
Inclusion Criteria:

* Have no allergic conjunctivitis.
* Not be using any topical ocular medications.

Exclusion Criteria:

* Considered by the Investigator to not be a suitable candidate for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Specific characteristics are that one group will be habitual contact lens wearers, and the other group will be non-contact lens wearers (not having worn contact lenses within the last 7 days prior to baseline visit)
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Steffen, OD, MS, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Incorporated, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Contact Lens Wear | Non-Contact Lens Wear
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Contact Lens Wear | Non-Contact Lens Wear | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Median (Full Range); unit: years] | 41 [23 to 59] | 41 [29 to 49] | 41 [23 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Hyaluronan Levels
Description: Tear samples collected using a Schirmer tear strip and analyzed for hyaluronan (HA) levels, a lubricant found throughout the body, including tears. Levels will be compared between the lens wearers and non-lens wearers.
Time Frame: 7 days following lens insertion
Population: DUE TO THE CANCELLATION OF THIS PROJECT, NO STATISTICAL OR CLINICALLY MEANINGFUL CONCLUSIONS RELATED TO THE STUDY ENDPOINTS WERE MADE.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Contact Lens Wear | Non-Contact Lens Wear
Number analyzed (Participants) | 12 | 13
ng/mL | 4.52 (.232) | 4.07 (.183)

ADVERSE EVENTS:
Arm/Group | Contact Lens Wear | Non-Contact Lens Wear
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes